CLINICAL TRIAL: NCT04941430
Title: Pilot Study of 7T MRI for Early Diagnosis of Melanoma Brain Metastases
Brief Title: 7T MRI Scan for the Early Detection of Melanoma Brain Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10M-20-1; NCI-2021-05850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10M-20-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (7T MRI) (Experimental): Within 2 weeks of initial standard of care 3T MRI, patients undergo 7T MRI scan with and without contrast over 1-2 hours.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging using 7 Tesla MRI

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging using 7 Tesla MRI — Undergo 7T MRI
  Other Names: 7 Tesla MRI; 7T MRI

SUMMARY:
This clinical trial studies the use of 7-Tesla (7T) magnetic resonance imaging (MRI) in detecting melanoma that has spread to the brain (melanoma brain metastases). The standard MRI brain imaging is done on 3T or similar MRI machine, but the 7T MRI machine has a larger magnet which has been shown to have superior resolution of the brain and of non-cancerous brain lesions. Diagnostic procedures such as 7T MRI may help find and diagnose melanoma brain metastases earlier than standard 3T MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the potential superiority of contrast-enhanced (CE) 7T MRI by comparing to standard of care CE 3T MRI in detecting occult brain metastases lesion at time of diagnosis of new brain metastases.

SECONDARY OBJECTIVE:

I. Describe the imaging characteristics of melanoma brain metastases on 7T MRI of the brain.

EXPLORATORY OBJECTIVE:

I. Evaluate incidence of diagnosis of leptomeningeal disease on CE 7T MRI brain.

OUTLINE:

Within 2 weeks of initial standard of care 3T MRI, patients undergo 7T MRI scan with and without contrast over 1-2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma patients with new untreated brain metastases seen on CE 3T MRI
* Patient may have received previous systemic therapy, immunotherapy, or checkpoint inhibitors
* Patient may have previous brain metastases treated >30 days prior with brain radiation, either whole brain radiation or radiosurgery
* Age >= 18 years
* Karnofsky performance status (KPS) >= 70
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of child-bearing potential need negative urine human chorionic gonadotropin (hCG) within 2 weeks prior to any treatment. A female of child-bearing potential is defined as any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to tolerate MRI (able to lie flat in supine position without undue anxiety or discomfort or history of claustrophobia)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have had brain neurosurgery =< 30 days prior to entering the study or those who have not recovered from adverse events related to that procedure
* Patients who have had central nervous system (CNS)-directed radiotherapy =< 30 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 30 days earlier
* Patients with claustrophobia or anxiety limiting ability to tolerate MRI scans. Unable to tolerate MRI scan without use of anxiolytic medication or with distress requiring termination of scan or resulting in scans of poor quality
* Patients with MRI-incompatible pacemakers or MRI-incompatible implants
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gadolinium-based contrast agents (GBCA) or other agents used in study
* Patients with poor renal function (estimated glomerular filtration rate [eGFR] < 30) or requiring dialysis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Presence or absence of brain metastases on 7 tesla (T) magnetic resonance imaging (MRI) as compared to the standard of care 3T MRI | Up to 14 days
  Any visualized brain metastases seen in this study on 3T will be evaluated using the criteria proposed by the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM). As there are no consensus criteria for 7T MRI published at this time, we will apply the same RANO-BM criteria to the study 7T MRI exams.Will count the discordant lesions between 3T and 7T, i.e. lesion identified in 7T but not 3T (L71L30) versus (vs.) lesion identified in 3T but not 7T(L70L31). McNemar's test will be used to compare L71L30 vs. L70L31. Will report 95% Clopper Pearson exact confidence interval for L71L30 vs. L70L31 in incidence of diagnosis of leptomeningeal disease.
Primary tumor size | Up to 14 days
  Measured by study contrast enhanced (CE) 7T MRI compared to standard of care 3T MRI.

OTHER OUTCOMES:
Incidence of diagnosis of leptomeningeal disease on CE 7T MRI brain | At baseline
  Spaghetti plots will be used to illustrate the radiographic patterns of unique tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Hwang, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States